CLINICAL TRIAL: NCT01461005
Title: A Postmarket Surveillance Study of the Paradigm Spine Dynamic Stabilization System(DSS)
Brief Title: A Postmarket Surveillance Study of the Paradigm Spine Dynamic Stabilization System (DSS)
Acronym: DSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA reclassified so all 522 studies were stopped,
Sponsor: Paradigm Spine (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dynamic Stabilization System
Record Dates: First submitted 2011-10-18; First posted 2011-10-27 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Spondylolisthesis; Neurologic Deficits; Kyphosis; Pseudarthrosis
Keywords: Spondylolisthesis; Neurologic impairment; Kyphosis; Pseudarthrosis
MeSH Terms: conditions — Spondylolisthesis; Neurologic Manifestations; Kyphosis; Pseudarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dynamic Stabilization System (Experimental): Dynamic Stabilization System (DSS) System
  Interventions: Device: Dynamic Stabilization System (DSS)

INTERVENTIONS:
Device: Dynamic Stabilization System (DSS) — Dynamic Stabilization System

SUMMARY:
The purpose of the Post-Market Surveillance study is to evaluate safety.

DETAILED DESCRIPTION:
Paradigm Spine Dynamic Stabilization System (DSS) study is a prospective, multi-center, literature controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature (21-85 years old).
* Patient has degenerative spondylolisthesis (Grade 1-3) with objective evidence of neurologic impairment, kyphosis, and/or failed previous fusion (pseudarthrosis) at index level.
* Capable and willing to comply with the requirements unique to the study, adhere to the post-operative treatment and management program, and return for required follow-up examinations.
* Surgeon has determined that DSS™ System is an appropriate treatment for the patient without regard to the study.

Exclusion Criteria:

* The need for interbody cages, allograft, or any other assistance during surgery. Device is only to be used with autograft per FDA approved indications.
* Any medical, mental or surgical condition precluding the potential benefit of spinal surgery or surgery in general.
* Acute or chronic systemic, spinal or localized infections.
* Active, severe systemic and metabolic diseases.
* Obesity defined as Body Mass Index > 35.
* Subject is pregnant or interested in becoming pregnant in the next 36 months.
* Dependency on pharmaceutical drugs, drug abuse, or alcoholism.
* Lack of patient cooperation.
* Foreign body sensitivity to the implant material.
* Degenerative scoliosis greater than 25 degrees.
* Grade 4 degenerative spondylolisthesis (>75% slip).
* Significant osteopenia A screening questionnaire for osteopenia, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a DEXA bone mineral density measurement. If DEXA is required*, exclusion will be defined as a DEXA bone density measured T score of ≤ -1.0 (The World Health Organization definition of osteopenia).
* Soft tissue deficit not allowing wound closure.
* Congenital abnormalities, tumors or other conditions that would prevent secure component fixation that has the potential to decrease the useful life of the device.
* Inadequate pedicles or vertebral body geometry of the thoracic, lumbar and sacral vertebrae.
* Bony lumbar spinal stenosis not related to the primary degenerative spondylolisthesis indication.
* Pars defect.
* Clinically compromised vertebral bodies at affected level due to current or past trauma.
* Prisoner or ward of the state.
* Currently in litigation regarding a spinal condition.
* Known allergy to titanium, titanium alloys, CoCrMo, polyethylene or MR contrast agents.
* Is currently involved in a study of another investigational product for similar purpose.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitela Gandelman, Study Director — Paradigm Spine LLC
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dynamic Stabilization System
Started | 1
Completed | 0
Not Completed | 1
Not completed — FDA reclassified Dynamic Stabilization D | 1

BASELINE CHARACTERISTICS:
Groups:
- DSS Stabilization System: DSS Stabilization System
Arm/Group | DSS Stabilization System
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have an Incidence of Serious or Device Related Adverse Events Due to Device or Procedure.
Description: The safety endpoint is defined as the incidence of serious or device related adverse events attributable to the device or procedure. Reoperations, revisions or removals of the Dynamic Stabilization System (DSS) System implant will be evaluated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Stabilization System
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Measurement of Lower Back Pain as Assessed by Visual Analog Scale
Description: Lower back pain as measured by the Visual Analog Scale (VAS) on the scale from 0 (no pain) to 100 (worst imaginable pain)
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | Dynamic Stabilization System
Number analyzed (Participants) | 1
units on a scale | 2

3. Secondary Outcome: Measurement of Right Leg Pain as Assessed by Visual Analog Scale
Description: Right leg pain as measured by the Visual Analog Scale (VAS) on the scale from 0 (no pain) to 100 (worst imaginable pain)
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | DSS Stabilization System
Number analyzed (Participants) | 1
units on a scale | 2

4. Secondary Outcome: Measurement of Left Leg Pain as Assessed by Visual Analog Scale
Description: Left leg pain as measured by the Visual Analog Scale (VAS) on the scale from 0 (no pain) to 100 (worst imaginable pain)
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | DSS Stabilization System
Number analyzed (Participants) | 1
units on a scale | 12

5. Secondary Outcome: Number of Participants With Improved Health as Measured by the EuroQOL Health Related Qualify of Life- 5 Dimensions-3 Level (EQ-5D-3L) Health Questionnaire Compared to Baseline.
Description: The EQ-5D-3L is a standardized instrument used as a measure of health outcomes. It contains questions in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and provides a simple descriptive profile and single index for health status preference. In addition, there is a Visual Analog Scale (VAS). The VAS is the participant's rating of their health on a scale of 0 "worst imaginable health state" to 100 "best imaginable health state".
Time Frame: Pre-Op, 6 weeks, 6 months, 12 months, and 24 months
Measure: Number; unit: participants
Arm/Group | DSS Stabilization System
Number analyzed (Participants) | 1
participants | 1

6. Secondary Outcome: Assessment of Back Pain Using the Oswestry Low Back Pain Disability Index (ODI).
Description: ODI is a questionnaire that provides information on back and the affects on managing every day life by diving questions into 10 sections. The total possible score for each section is 0-5. The scores are then converted into percentages ranging from 0% (minimal disability) to 100% (maximum possible disability).
Time Frame: 6 months
Measure: Number; unit: score on a scale
Arm/Group | DSS Stabilization System
Number analyzed (Participants) | 1
score on a scale | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Dynamic Stabilization System
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days